CLINICAL TRIAL: NCT05302076
Title: Evaluation the Effect of Low-intensity Electrical Current (LIEC) in Accelerating the En-masse Retraction of the Maxillary Anterior Teeth and the Associated Skeletal, Dental and Periodontal Changes : A Randomized Controlled Clinical Trial
Brief Title: Clinical Effects of Electrical Stimulation on Speeding up Orthodontic Tooth Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-05-2022
Record Dates: First submitted 2022-03-20; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Class II Malocclusion
Keywords: En-masse retraction; Acceleration; Low-intensity electric current
MeSH Terms: conditions — Overbite

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electric current (Experimental): Electric current will be applied in this group of patients using removable device.
  Interventions: Device: Low-intensity electrical current (LIEC)
- Traditional treatment (Active Comparator): No acceleration method will be performed in this group.
  Interventions: Device: Traditional fixed orthodontic appliance

INTERVENTIONS:
Device: Low-intensity electrical current (LIEC) — Each patient in the electrical group will be asked to wear a removable device containing a small electrical circuit that will supply the required electric current for five hours a day until the completion the retraction of the upper anterior teeth.
  Arms: electric current
Device: Traditional fixed orthodontic appliance — The maxillary arch will be levelled and aligned. The rectangular stainless steel archwires (0.019" × 0.025") with anterior 8mm height soldered hooks distal to the canines will be inserted. (250-300) g force will be applied on each side using two NiTi springs attached between the mini-implants and the soldered hooks in a direction approximately parallel to the occlusal plane for conducting an en-masse retraction.
  Arms: Traditional treatment

SUMMARY:
Thirty two patients requiring extraction of maxillary first premolars and en-masse retraction of upper anterior teeth will participate in the study. They will be divided randomly into two groups: electrical group and control group. In each group, en-masse retraction will be initiated after completion of the leveling and alignment phase via closed nickel-titanium coil springs applying 250 g of force per side, Mini-implants will be used as an anchor unit.

The overall retraction duration will be calculated. The skeletal, dental and soft tissue changes will be detected using panoramic and lateral cephalometric radiographs which will be obtained pretreatment, pre and post en-masse retraction of the anterior teeth.

DETAILED DESCRIPTION:
Prior to enrollment of each subject into the study, they will be examined completely to determine the orthodontic treatment plan. The operator will inform them about the aim of the study and ask them to provide a written informed consent.

Self-drilling titanium mini-implants (1.6mm diameter and 8mm length) will be used. They will be inserted between the maxillary second premolar and first molar at approximately 8-10 mm above the archwires at the mucogingival junction and will be checked for primary stability (mechanical retention). Then the maxillary first premolar will be extracted. The maxillary arch will be levelled and aligned. The rectangular stainless steel archwires (0.019" × 0.025") with anterior 8mm height soldered hooks distal to the canines will be inserted.

A removable device containing a small electrical circuit will be applied to each patient to supply the required electric current.

Each patient in the electrical group will be asked to wear a removable device containing a small electrical circuit that will supply the required electric current for five hours a day until the completion the retraction of the upper anterior teeth.

(250-300) g force will be applied on each side using two NiTi springs attached between the mini-implants and the soldered hooks in a direction approximately parallel to the occlusal plane for conducting an en-masse retraction. The force level will be measured every 2 weeks. Retraction will be stopped when a class I canine relationship will be achieved and a good incisor relationship will be obtained.

The duration of retraction will be calculated by calculating the time required to achieve complete retraction of the upper anterior teeth through clinical examination.

Panoramic and lateral cephalometric radiographs will be obtained pretreatment, pre and post en-masse retraction of the anterior teeth, to assess the skeletal, dental and soft tissue changes.

Periodontal health will be assessed at the beginning of orthodontic treatment, before and after en-masse retraction by evaluating the following parameters: plaque index, gingival index, bleeding index, probing depth and gingival recession.

ELIGIBILITY:
Inclusion Criteria:

1. Adult healthy patients, Male and female, Age range: 15-27 years.
2. Class II Division 1 malocclusion :

   * Mild / moderate skeletal Class II (sagittal discrepancy angle ≤7)
   * Overjet ≤10
   * Normal or excessive facial height (Clinically and then cephalometrically assessed using these three angles : mandibular/cranial base angle, maxillary/mandibular plane angle and facial axis angle)
   * Mild to moderate crowding ≤ 4
3. Permanent occlusion.
4. Existence of all the upper teeth (except third molars).
5. Good oral and periodontal health:

   * Probing depth < 4 mm
   * No radiographic evidence of bone loss.
   * Gingival index ≤ 1
   * Plaque index ≤ 1

Exclusion Criteria:

1. Medical problems that affect tooth movement (corticosteroid, nonsteroidal anti-inflammatory drugs (NSAIDs), …)
2. Presence of primary teeth in the maxillary arch
3. Missing permanent maxillary teeth (except third molars).
4. Poor oral hygiene or Current periodontal disease:

   * Probing depth ≥ 4 mm
   * radiographic evidence of bone loss
   * Gingival index > 1
   * Plaque index > 1
5. Patient had previous orthodontic treatment

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-12-05 (Actual)

PRIMARY OUTCOMES:
Duration of en-masse retraction of anterior teeth | The months required to complete the retraction procedure will be recorded. Completion of this procedure is expected to be occur within six months in the experimental group and eight months in the control group.
  Assessment will be performed by calculating the time required to achieve complete retraction of the upper anterior teeth (six teeth) through clinical examination.
Change in the SN-U1 angle | : The cephalogram will be taken twice, 1 week before the commencement of the retraction and at the completion of retraction. Completion of this procedure is expected to be done within 6 months in the experimental group and 8 months in the control group.
  This angle the represents the relationship of the upper anterior teeth with SN in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken and this angle is going to be measured in degrees.
Change in the SNA angle | : The cephalogram will be taken twice, 1 week before the commencement of the retraction and at the completion of retraction. Completion of this procedure is expected to be done within 6 months in the experimental group and 8 months in the control group.
  This angle the represents the position of the upper jaw in the cephalometric analysis in the anteroposterior direction. Lateral cephalograms will be taken and this angle is going to be measured in degrees.
Change in the MM angle | : The cephalogram will be taken twice, 1 week before the commencement of the retraction and at the completion of retraction. Completion of this procedure is expected to be done within 6 months in the experimental group and 8 months in the control group.
  This angle the represents the amount of vertical divergence between the upper and lower jaws in the cephalometric analysis. Lateral cephalograms will be taken and this angle is going to be measured in degrees.

SECONDARY OUTCOMES:
Change in the Nasolabial angle | : The cephalogram will be taken twice, 1 week before the commencement of the retraction and at the completion of retraction. Completion of this procedure is expected to be done within 6 months in the experimental group and 8 months in the control group.
  This angle the represents the relationship of the upper lip with nose in the cephalometric analysis. Lateral cephalograms will be taken and this angle is going to be measured in degrees.
Change in the Li-E Line | : The cephalogram will be taken twice, 1 week before the commencement of the retraction and at the completion of retraction. Completion of this procedure is expected to be done within 6 months in the experimental group and 8 months in the control group.
  This measurement represents the relationship between the upper lip and the Ricketts line in cephalometric analysis. Lateral cephalograms will be taken and this variable will be measured in mm.
Change in Root Length | This will be measured: one day before the commencement of the retraction phase and at the end of the retraction phase which is expected to occur within 6 months in the experimental group and 8 months in the control group.
  The root length will be measured for each root of six upper anterior teeth using panorama imaging, the change will be calculated between before and after images in mm.
Change in the Plaque index | This will be measured: one day before the commencement of the retraction phase and at the end of the retraction phase which is expected to occur within 6 months in the experimental group and 8 months in the control group.
  The plaque index will be used to assess the status of the oral hygiene in these patients.
Change in the Gingival Index | This will be measured: one day before the commencement of the retraction phase and at the end of the retraction phase which is expected to occur within 6 months in the experimental group and 8 months in the control group.
  The Gingival index will be used to assess the status of the gingival tissues around the teeth.
Change in the Bleeding Index | This will be measured: one day before the commencement of the retraction phase and at the end of the retraction phase which is expected to occur within 6 months in the experimental group and 8 months in the control group.
  The Bleeding index will be used to assess the status of periodontal tissues and the amount of congestion in the gingival margins around the anterior teeth.
Change in the Probing Depth | Two measurements are required for this calculation: one day before the commencement of the retraction phase and at the end of the retraction phase which is expected to occur within 6 months in the experimental group and 8 months in the control group.
  This will be measured in millimeters from the gingival margin to the bottom of the sulcus/pocket around the six anterior teeth.
Change in the Gingival Recession | Two measurements are required for this calculation: one day before the commencement of the retraction phase and at the end of the retraction phase which is expected to occur within 6 months in the experimental group and 8 months in the control group.
  This will be measured in millimeters from the cement-enamel junction to the level of the gingival margin around the six anterior teeth.

CONTACTS AND LOCATIONS:
Overall Officials: Rashad Ibrahem Shaadouh, DDS, Principal Investigator — Department of orthodontics, Damascus University, Syria; Mohammad Y Hajeer, DDS,MSc,PhD, Study Director — Department of orthodontics, Damascus University, Syria; Ghiath Mahmoud, DDS,MSc,PhD, Study Director — Department of orthodontics, Damascus University, Syria
Locations (1):
- University of Damascus, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davidovitch Z, Finkelson MD, Steigman S, Shanfeld JL, Montgomery PC, Korostoff E. Electric currents, bone remodeling, and orthodontic tooth movement. II. Increase in rate of tooth movement and periodontal cyclic nucleotide levels by combined force and electric current. Am J Orthod. 1980 Jan;77(1):33-47. doi: 10.1016/0002-9416(80)90222-5. PMID 6243448
- [Background] Spadari GS, Zaniboni E, Vedovello SA, Santamaria MP, do Amaral ME, Dos Santos GM, Esquisatto MA, Mendonca FA, Santamaria M Jr. Electrical stimulation enhances tissue reorganization during orthodontic tooth movement in rats. Clin Oral Investig. 2017 Jan;21(1):111-120. doi: 10.1007/s00784-016-1759-6. Epub 2016 Feb 26. PMID 26917494
- [Background] Zaniboni E, Bagne L, Camargo T, do Amaral MEC, Felonato M, de Andrade TAM, Dos Santos GMT, Caetano GF, Esquisatto MAM, Santamaria M Jr, Mendonca FAS. Do electrical current and laser therapies improve bone remodeling during an orthodontic treatment with corticotomy? Clin Oral Investig. 2019 Nov;23(11):4083-4097. doi: 10.1007/s00784-019-02845-9. Epub 2019 Feb 15. PMID 30771000
- [Background] Chaudhari SD, Sharma KK, Marchetto JJ, Hydren JR, Burton BM, Moreno AP. Modulating OPG and TGF-beta1 mRNA expression via bioelectrical stimulation. Bone Rep. 2021 Oct 9;15:101141. doi: 10.1016/j.bonr.2021.101141. eCollection 2021 Dec. PMID 34692946
- [Background] Gkantidis N, Mistakidis I, Kouskoura T, Pandis N. Effectiveness of non-conventional methods for accelerated orthodontic tooth movement: a systematic review and meta-analysis. J Dent. 2014 Oct;42(10):1300-19. doi: 10.1016/j.jdent.2014.07.013. Epub 2014 Jul 27. PMID 25072362
- [Background] Masella RS, Meister M. Current concepts in the biology of orthodontic tooth movement. Am J Orthod Dentofacial Orthop. 2006 Apr;129(4):458-68. doi: 10.1016/j.ajodo.2005.12.013. PMID 16627170